CLINICAL TRIAL: NCT04882748
Title: Using a Robot to Treat Non-specific Low Back Pain: a Two-arm, Single-blinded, Randomized Controlled Trial
Brief Title: Using a Robot to Treat Non-specific Low Back Pain
Acronym: ADAMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Rioja Salud (Other)
Collaborators: Hospital San Pedro de Logroño (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRS-ADAMO-01
Record Dates: First submitted 2021-04-29; First posted 2021-05-12 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Non-specific Low Back Pain
Keywords: back pain; massage; robot
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Forty-four patients suffering from NSLBP will be recruited after signing the informed consent and randomly assigned to one of two experimental arms: physical therapy with or without the help of a robot for 10 sessions. Pain evaluation will be performed with the Oswestry disability index (ODI), which will be applied before starting and at the end of the treatment, and the visual analogue scale (VAS) which will be applied after each session. The ODI will be performed by an independent physician blind to the treatment. Statistical analysis will be performed to compare both treatments.
Who Masked: Outcomes Assessor
Masking Description: The Oswestry disability index (ODI) will be performed by an independent physician blind to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): In the control arm, patients were laid down on the robot platform. Physiotherapists identified the trigger points and the robot was connected, providing the expected noise and vibration, but the air pressure was not applied. Thermotherapy and rehabilitation exercises were provided, as is the standard treatment for NSLBP at the Rehabilitation Service.
  Interventions: Other: ADAMO
- Robot massage (Experimental): In the robot arm, a physiotherapist with more than 15 years of experience identified the trigger points in the patient, programmed the robot, and applied robot-controlled air pressure massage for 10 minutes. The ADAMO robot applies an air current to the trigger points on the back of the patient, guided by cameras and computer programs (https://adamorobot.com/). Thermotherapy and rehabilitation exercises were also applied.
  Interventions: Other: ADAMO

INTERVENTIONS:
Other: ADAMO — Physical therapy provided with or without the help of a robot

SUMMARY:
Non-specific low back pain (NSLBP) is a musculoskeletal syndrome whose main characteristic is the pain, which is focalized in the lumbar area of the spine, which cannot be attributed to a known cause (traumatism, systemic diseases, nerve root compression, etc). The treatment includes massage and rehabilitation techniques. Here the investigators want to test whether a robot (ADAMO) may help in improving current physiotherapy exercises in reducing back pain. NSLBP patients will be randomly assigned to two arms (robot versus control) and they will receive 10 massage sessions. Pain evaluation will be performed with the visual analogue scale (VAS) and the Oswestry disability index (ODI). The ODI will be performed by an independent physician blind to the treatment.

DETAILED DESCRIPTION:
Low back pain is defined as a musculoskeletal syndrome, or group of symptoms, whose main characteristic is the pain, which is focalized in the lumbar area of the spine. The diagnosis is rather easy since symptoms are very evident. When this pain cannot be attributed to a known cause (traumatism, systemic diseases, nerve root compression, etc), it is called non-specific low back pain (NSLBP), which may represent 90-95% of all cases of back pain.

The treatment for this pathology has been collected in several clinical practice guidelines, with little differences among them. All of them recommend: i) maintaining physical activity as far as the pain allows; ii) pharmacological treatment (analgesics, non-steroidal anti-inflammatories, muscle relaxants); and iii) non-pharmacological measures (local heat, cognitive-behavior therapy, spinal manipulation, rehabilitation programs). Rehabilitation therapy, including different exercises, such as extensions, back workshops, and aquatic exercises, among others, provides excellent results in managing chronic back pain. In addition, physiotherapeutic massage constitutes the most common practice to treat back pain and is very effective in the short term, although it may not address the underlying causes.

The main problem in reporting and measuring physiotherapeutic massage practices is that the massage is applied by different therapists, with different strength and intensity, which may vary from session to session. The use of massaging robotic devices should solve all these problems and several prototypes are already available.

In this study, the efficiency of the new ADAMO robot system (https://adamorobot.com/) will be tested. ADAMO bases its operation on a computer program that controls the manipulator robot, which, and by means of cameras installed at its end, must find in each session the points of treatment in the patient previously defined by the health professional and apply the air at the necessary pressure. This pressure is generated by means of a compressed air nozzle integrated in a handpiece installed at the end of the robot.

Forty-four patients suffering from NSLBP will be recruited after signing the informed consent and randomly assigned to one of two experimental arms: robot or control for 10 sessions. Pain evaluation will be performed with the Oswestry disability index (ODI), which will be applied before starting and at the end of the treatment, and the visual analogue scale (VAS) which will be applied after each session. The ODI will be performed by an independent physician blind to the treatment. Statistical analysis will be performed to compare both treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering non-specific low back pain

Exclusion Criteria:

* Age <18 or >60 years Pregnant women Impossibility to stay in a prone position Serious systemic pathologies Patients with treatments that may interfere with the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Patient disability as tested by the Oswestry disability index (ODI). | Through study completion. An average of 6 months.
  The ODI will be recorded before starting and at the end of the treatment. The Oswestry disability index (ODI) is a questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. Possible scores go from 0 to 50, being 0 no pain and 50 the highest possible pain.
Perceived pain as tested by the visual analogue scale (VAS). | Through study completion. An average of 6 months.
  The VAS will be recorded after every session. The visual analogue scale (VAS) is a unidimensional measure of pain intensity. The patient is presented with a horizontal line of face pictograms. The patient marks on the line the point that they feel represents their perception of their current state, which may rank from 0 (best, no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Mirpuri, PhD, Study Director — CIBIR
Locations (1):
- CIBIR, Logroño, La Rioja, Spain

IPD SHARING:
Plan to Share IPD: Yes
All results from the study will be published in a specialized journal, including the study protocol, statistical Analysis, informed consent form, and a table with all raw data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be published together with the actual publication.
Access Criteria: Everyone will be able to access all data.

REFERENCES:
- [Result] Marin-Mendez H, Marin-Novoa P, Jimenez-Marin S, Isidoro-Garijo I, Ramos-Martinez M, Bobadilla M, Mirpuri E, Martinez A. Using a Robot to Treat Non-specific Low Back Pain: Results From a Two-Arm, Single-Blinded, Randomized Controlled Trial. Front Neurorobot. 2021 Sep 14;15:715632. doi: 10.3389/fnbot.2021.715632. eCollection 2021. PMID 34594197
- See also: Robot description — https://adamorobot.com/
- Available data/document: Individual Participant Data Set — https://www.frontiersin.org/articles/10.3389/fnbot.2021.715632/full#supplementary-material